CLINICAL TRIAL: NCT06468514
Title: Effectiveness of 'Tensioning Techniques' vs 'Sliding Techniques' on Radial Nerve for the Treatment of Lateral Epicondylalgia
Brief Title: Effectiveness of Neurodinamic Techniques on Radial Nerve for the Treatment of Lateral Epicondylalgia
Acronym: TT-ST-RN-LE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, MARIA BALSA AMARANTE, PT, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TECHNIQUES ON RADIAL NERVE
Record Dates: First submitted 2024-06-15; First posted 2024-06-21 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Epicondylalgia Neural mobilization Neural tension Physiotherapy Radial nerve
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRUPO 1 (Experimental): a Neural tension technique on the radial nerve will be performed.
  Interventions: Other: neural tensioning technique on radial nerve
- GRUPO 2 (Experimental): A neural gliding technique will be performed on the radial nerve.
  Interventions: Other: Sliding technique on radial nerve

INTERVENTIONS:
Other: neural tensioning technique on radial nerve — the neural group tensioning technique: The test should be performed in approximately 10° of shoulder abduction. The examiner extends the elbow 2 seconds just to the range where the patient notices tension but no pain and then the elbow is flexed. Three sets of 6-8 swings are performed with 1 minute rest in between.
  Arms: GRUPO 1
Other: Sliding technique on radial nerve — The mobilization maneuver begins by identifying the first resistance and the range of extension associated with pain. Maintaining elbow extension within the elastic region of resistance free of pain and/or paresthesia the examiner increases elbow extension and simultaneously allows the wrist to extend as necessary for the radial nerve branches in the forearm to glide proximally. The physical therapist then flexes the wrist while allowing the elbow to flex to cause the radial nerve excursion distally in the forearm.
  Arms: GRUPO 2

SUMMARY:
Lateral elbow pain is a prevalent musculoskeletal disorder in the working population due to overuse of the upper limb. This pathology has serious consequences for health, work performance and overall health burden.

In this injury, as in any musculoskeletal disorder, the peripheral nervous system is involved. Because of its course and corresponding motor and sensory innervation in the area, the radial nerve should be taken into consideration as a structure involved in elbow pain.

The aim of the present study is to demonstrate which of the neurodynamic techniques is more effective in lateral epicondylalgia, neural tension techniques or neural mobilization techniques.

DETAILED DESCRIPTION:
The aim of the present study is to demonstrate which is more effective among the neurodynamic techniques for lateral epicondylalgia, neural tension techniques or neural mobilization techniques.

A total of 60 subjects will be recruited and divided into 2 groups. 30 in Group 1 where they will receive a neural mobilization technique on the radial nerve and 30 in Group 2 where they will be subjected to a neural tension technique on the radial nerve.

The data to be collected will be grip strength, pain on pressure, pain and quality of life dash questionnaire, these data will be measured pre, post treatment and a re-evaluation at 4 weeks and 24 weeks after the intervention.

The duration of the treatment is 6 weeks, performing two sessions per week with 72 hours of rest between sessions. A total of 12 sessions will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with lateral epicondylalgia.
* Experiencing elbow pain of 2 to 6 months duration.
* Age between 30 and 60 years old.
* Radial humeral joint tenderness to palpation.
* Positive Cozen's test

Exclusion Criteria:

* - Bilateral symptoms.
* Rheumatologic disease involving the elbow and wrist
* Musculoskeletal disorder due to connective tissue pathology
* Cervical radiculopathy
* Nerve compression including the upper extremity
* Operation on the affected arm
* Having received treatment for epicondylalgia in the last 6 months
* Radiating pain from the cervical spine
* Instability of the external ligamentous complex of the elbow(3).
* Not having received any physiotherapy session in the month prior to the start of the study.
* Neural clinical manifestations (electric shock-like pain, tingling, tingling, numbness and/or burning).

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2025-03-24 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Grip strength | the duration of the program will be 6 weeks, with two sessions per week with 72 hours of rest between sessions. A total of 12 sessions will be carried out. A re-evaluation will be done 4 weeks after the final evaluation and another one after 24 weeks.
  his is a continuous quantitative variable. The measurement of grip strength is performed with the subject in a chair with backrest and armrests, his shoulder is in neutral position, and in adduction; the elbow in 90º flexion and the wrist in 30º extension. Participants are asked to perform maximal grip strength with the dynamometer in a self-selected grip position for 6 seconds. According to the American Society of Hand Therapists Guide, a Jamar® hydraulic dynamometer (Lafayette Instrument Company, USA) is used. The measurements were repeated 3 times, with an interval of 1 minute and the mean of the 3 measurements was used for statistical analysis.

SECONDARY OUTCOMES:
Pain on pressure | the duration of the program will be 6 weeks, with two sessions per week with 72 hours of rest between sessions. A total of 12 sessions will be carried out. A re-evaluation will be done 4 weeks after the final evaluation and another one after 24 weeks.
  This is a continuous quantitative variable. The pain threshold to pressure at the lateral epicondyle was measured with an algometer. The subject remains seated with the arm in 30° of abduction; the elbow in 90° of flexion; and with the forearm, wrist and hand resting on a table. The investigating physical therapist lightly palpates the common extensor tendon to identify the most tender area. Then, starting on the unaffected side, the head of the algometer (hard rubber tip, 1 cm2 surface area) is placed perpendicular to the common extensor tendon at the lateral epicondyle until the patient indicates the moment when the pressure sensation changes to pain. Three measurements are taken on both sides, with a 20-second rest interval between each measurement. The intraobserver reliability of these 3 measurements was excellent (ICC range, .91-.96). For the analysis, the mean value (in kg/cm2 ) of the 3 stresses was calculated. The maximum applied pressure was 6 kg/cm2 .
global pain | the duration of the program will be 6 weeks, with two sessions per week with 72 hours of rest between sessions. A total of 12 sessions will be carried out. A re-evaluation will be done 4 weeks after the final evaluation and another one after 24 weeks.
  This is a discrete quantitative variable. Pain was measured using the Numerical Pain Rating Scale (NRS-P). The procedure is as follows, the patient is asked at the present moment what pain he/she feels from 0 to 10 if zero is zero pain and 10 is the maximum pain he/she has perceived. The NRS-P is a 10 cm long line calibrated from 0 to 10. 10. The NRS has been shown to have a test-retest reliability of 0.64 to 0.86, from good to excellent (7).
DASH QUESTIONARY | the duration of the program will be 6 weeks, with two sessions per week with 72 hours of rest between sessions. A total of 12 sessions will be carried out. A re-evaluation will be done 4 weeks after the final evaluation and another one after 24 weeks.
  It is a discrete quantitative variable. The DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire is a self-administered outcome questionnaire that measures physical disability and symptoms of all upper extremity disorders. It includes 30 items related to 120 symptoms and activities of daily living. The total score is 100, and a higher score indicates a greater degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: María Balsa-Amarante, MSc, Principal Investigator — University of Alcalá
Locations (1):
- Campus Científico Tecnológico. Av. de León. 3A, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gamelas T, Fernandes A, Magalhaes I, Ferreira M, Machado S, Silva AG. Neural gliding versus neural tensioning: Effects on heat and cold thresholds, pain thresholds and hand grip strength in asymptomatic individuals. J Bodyw Mov Ther. 2019 Oct;23(4):799-804. doi: 10.1016/j.jbmt.2019.04.011. Epub 2019 Apr 24. PMID 31733764
- [Background] Ellis R, Carta G, Andrade RJ, Coppieters MW. Neurodynamics: is tension contentious? J Man Manip Ther. 2022 Feb;30(1):3-12. doi: 10.1080/10669817.2021.2001736. Epub 2021 Nov 16. PMID 34781843
- [Background] Yilmaz K, Yigiter Bayramlar K, Ayhan C, Tufekci O. Investigating the effects of neuromobilization in lateral epicondylitis. J Hand Ther. 2022 Jan-Mar;35(1):97-106. doi: 10.1016/j.jht.2020.11.003. Epub 2020 Nov 13. PMID 33563509
- [Background] Arumugam V, Selvam S, MacDermid JC. Radial nerve mobilization reduces lateral elbow pain and provides short-term relief in computer users. Open Orthop J. 2014 Oct 17;8:368-71. doi: 10.2174/1874325001408010368. eCollection 2014. PMID 25352930
- [Background] Taylor A, Wolff AL. The forgotten radial nerve: A conceptual framework for treatment of lateral elbow pain. J Hand Ther. 2021 Apr-Jun;34(2):323-329. doi: 10.1016/j.jht.2021.05.009. Epub 2021 Jun 27. PMID 34193382